CLINICAL TRIAL: NCT00745264
Title: Multi-Centre, Open-Label, Two Segment, Parallel Group Study Comparing Plasma Pharmacokinetics of Ketoprofen in Diractin® Alone to Diractin® Applied Concomitant With Heat or Moderate Exercise
Brief Title: Multi-Centre, Open-Label, Two Segment, Study Comparing Plasma Pharmacokinetics of Ketoprofen in Diractin® Alone to Diractin® Applied Concomitant With Heat or Moderate Exercise
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IDEA AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CL-033-I-04
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Pharmacokinetic
Keywords: heat; exercise
MeSH Terms: conditions — Motor Activity

ARMS (4):
- 2 (Experimental): 400 mg Ketoprofen from Diractin to 4 joints
  Interventions: Drug: Diractin
- 3 (Experimental): 100 and 400 mg Ketoprofen used concomittant with heat
  Interventions: Drug: Diractin
- 4 (Experimental): 100 and 400 mg Ketoprofen concomittant with moderate exercise
  Interventions: Drug: Diractin
- 1 (Experimental): 100 mg ketoprofen to 2 joints
  Interventions: Drug: Diractin

INTERVENTIONS:
Drug: Diractin — 100 mg Ketoprofen to 2 joints
  Arms: 1
Drug: Diractin — 400 mg ketoprofen to 4 joints
  Arms: 2
Drug: Diractin — 100 and 400 mg Ketoprofen used concomittant with heat
  Arms: 3
Drug: Diractin — 100 and 400 mg Ketoprofen concomittant with moderate exercise
  Arms: 4

SUMMARY:
* Comparison of the plasma PK after single use of 100 mg ketoprofen from Diractin®. 50 mg applied on 2 major joints to
* 400 mg ketoprofen from Diractin® (100 mg applied to 4 joints - overexposure)
* 100 mg and 400 mg ketoprofen from Diractin® used concomitant with heat application
* 100 mg and 400 mg ketoprofen from Diractin® used concomitant with moderate exercise

ELIGIBILITY:
Inclusion Criteria:

* All of the following criteria have to be met to include a subject in the study:

  * Understands nature and provision of the study
  * Have been informed about the study by the investigator and gave signed and dated informed consent prior to participation
  * Male and female subjects
  * Age 18-55 years
  * Subjects in good health as determined by the Investigator
  * Woman of childbearing potential using reliable methods of contraception with a low failure rate (i.e. less than 1% per year), e.g. implants, injectables, combined oral contraceptives, reliable intrauterine-devices, vasectomised/ infertile partner or surgically sterile (uterus removed or both tubes tied) or postmenopausal (at least 2 years without periods)

Exclusion Criteria:

* 4.2.1 General Exclusion Criteria

  * Investigator or any other team member involved directly or indirectly in the conduct of the clinical trial
  * Subjects who are inmates of psychiatric wards, prisons, or other state institutions
  * Participation in another clinical trial within the last 30 days
  * Not willing to refrain from exposing target areas after treatment to excessive ultraviolet light (solar radiation or solarium)
  * Pregnancy or lactation

4.2.2 Medical History Related Exclusion Criteria

* Known hypersensitivity or allergy (including photoallergy) to NSAID´s including ketoprofen, and ingredients used in pharmaceutical products
* Alcohol or drug abuse
* Malignancy within the past 2 years
* Skin lesions, dermatological diseases or tattoo in the treatment area
* Major surgery 3 months before enrolment
* Impaired haematopoesis and coagulation
* Gastric and duodenal ulcer and gastrointestinal bleedings
* Systemic lupus erythematodes, mixed connective tissue disease
* Major heart disease / uncontrolled hypertension
* Hepatic failure with ALT and/or AST > 2.0 ULN
* Renal failure with serum creatinine levels > 1.5 milligrams/deciliter (mg/dL)
* Varicosis, thrombophlebitis and other vascular disorders of the lower extremities
* Major traumatic lesions (e.g. fracture, tendon or muscle ruptures) of the musculo-sceletal system of the lower limbs
* HIV - Infection
* Blood donation one (1) month before screening and during study
* Hepatitis B and C
* Asthma bronchiale

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Egbert Seidel, MD, PhD, Principal Investigator — X-pert Med GmbH
Locations (2):
- Germany (2):
  - X-pert Med GmbH, Jena
  - ClinPharm Interantional GmbH, Leipzig